CLINICAL TRIAL: NCT00445965
Title: Phase II Study of Intrathecal I-3F8 in Patients With GD2-Expressing Central Nervous System and Leptomeningeal Neoplasms
Brief Title: Iodine I 131 Monoclonal Antibody 3F8 in Treating Patients With Central Nervous System Cancer or Leptomeningeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-122; MSKCC-05122
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-02

CONDITIONS: Brain and Central Nervous System Tumors; Intraocular Melanoma; Lung Cancer; Melanoma (Skin); Metastatic Cancer; Neuroblastoma; Ovarian Cancer; Retinoblastoma; Sarcoma; Small Intestine Cancer
Keywords: recurrent childhood medulloblastoma; untreated childhood medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); recurrent childhood supratentorial primitive neuroectodermal tumor; untreated childhood supratentorial primitive neuroectodermal tumor; adult anaplastic astrocytoma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult subependymal giant cell astrocytoma; recurrent childhood subependymal giant cell astrocytoma; untreated childhood subependymal giant cell astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; untreated childhood cerebellar astrocytoma; adult brain stem glioma; adult mixed glioma; childhood mixed glioma; recurrent childhood brain stem glioma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway glioma; untreated childhood brain stem glioma; untreated childhood visual pathway and hypothalamic glioma; untreated childhood visual pathway glioma; regional neuroblastoma; disseminated neuroblastoma; recurrent neuroblastoma; extraocular retinoblastoma; recurrent retinoblastoma; adult anaplastic ependymoma; adult ependymoblastoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent childhood ependymoma; childhood atypical teratoid/rhabdoid tumor; recurrent melanoma; stage IV melanoma; adult medulloblastoma; chondrosarcoma; metastatic osteosarcoma; recurrent osteosarcoma; metastatic childhood soft tissue sarcoma; ovarian sarcoma; recurrent childhood soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; previously treated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; adult anaplastic oligodendroglioma; adult desmoplastic small round cell tumor; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; tumors metastatic to brain; adult rhabdomyosarcoma; childhood oligodendroglioma; childhood desmoplastic small round cell tumor; extensive stage small cell lung cancer; intraocular retinoblastoma; recurrent adult brain tumor; recurrent adult soft tissue sarcoma; recurrent uterine sarcoma; small intestine leiomyosarcoma; recurrent small intestine cancer; recurrent small cell lung cancer; extraocular extension melanoma; recurrent intraocular melanoma; metastatic intraocular melanoma; iris melanoma; ciliary body and choroid melanoma, medium/large size; newly diagnosed childhood ependymoma; adult glioblastoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood pineoblastoma; untreated childhood pineoblastoma; adult pineal gland astrocytoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma; recurrent childhood anaplastic astrocytoma; untreated childhood anaplastic astrocytoma; recurrent childhood anaplastic oligoastrocytoma; recurrent childhood anaplastic oligodendroglioma; untreated childhood anaplastic oligoastrocytoma; untreated childhood anaplastic oligodendroglioma; recurrent childhood giant cell glioblastoma; recurrent childhood glioblastoma; untreated childhood giant cell glioblastoma; untreated childhood glioblastoma; recurrent childhood gliosarcoma; untreated childhood gliosarcoma; recurrent childhood gliomatosis cerebri; untreated childhood gliomatosis cerebri; childhood high-grade cerebellar astrocytoma; childhood high-grade cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Uveal Melanoma; Lung Neoplasms; Melanoma; Neoplasm Metastasis; Neuroblastoma; Ovarian Neoplasms; Retinoblastoma; Sarcoma; Medulloblastoma; Astrocytoma; Glioma; Optic Nerve Glioma; Ependymoma; Neuroectodermal Tumors, Primitive; Glioma, Subependymal; Familial ependymoma; Rhabdoid Tumor; Chondrosarcoma; Osteosarcoma; Oligodendroglioma; Desmoplastic Small Round Cell Tumor; Glioblastoma; Gliosarcoma; Brain Neoplasms; Rhabdomyosarcoma; Small Cell Lung Carcinoma; Neuroectodermal Tumors, Primitive, Peripheral; Neoplasms, Neuroepithelial | interventions — Immunologic Techniques

ARMS (1):
- 131I-3F8 (Experimental): This is a phase II single-arm open-label study that will define responses to therapy with weekly intrathecal 131I-3F8 in patients with central nervous system/leptomeningeal GD2-expressing disease.
  Interventions: Genetic: DNA analysis; Other: immunologic technique; Other: pharmacological study; Radiation: iodine I 131 monoclonal antibody 3F8; Radiation: 131I-3F8

INTERVENTIONS:
Genetic: DNA analysis
Other: immunologic technique
Other: pharmacological study
Radiation: iodine I 131 monoclonal antibody 3F8
Radiation: 131I-3F8 — Patients will receive 10mCi intrathecal 131I-3F8 per week. Patients will be pre-medicated with dexamethasone to prevent possible meningeal inflammatory reaction, Liothyronine and SSKI to prevent thyroid accumulation, and acetaminophen and diphenhydramine in anticipation of possible allergic reaction and fever.

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies, such as iodine I 131 monoclonal antibody 3F8, can find tumor cells and carry tumor-killing substances to them without harming normal cells. This may be an effective treatment for central nervous system cancer or leptomeningeal metastases.

PURPOSE: This phase II trial is studying the side effects and how well iodine I 131 monoclonal antibody 3F8 works in treating patients with central nervous system cancer or leptomeningeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if intrathecal iodine I 131 monoclonal antibody 3F8 activity in patients with GD2-expressing central nervous system or leptomeningeal neoplasms is sufficiently promising (i.e., 6-month overall survival rate ≥ 25%) to warrant further study.
* Determine the response rate in patients treated with this drug.
* Determine the cumulative toxicities of this drug in these patients.
* Describe the effects of human-antimouse antibody on cerebrospinal fluid and serum pharmacokinetics in patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive intrathecal iodine I 131 monoclonal antibody 3F8 for dosimetry. Beginning approximately 1 week later, patients receive intrathecal iodine I 131 monoclonal antibody 3F8 on day 1. Treatment intrathecal iodine I 131 monoclonal antibody 3F8 repeats weekly for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Blood and cerebrospinal fluid samples are collected prior to and after administration of each course of study drug. Samples are analyzed to assess the intrathecal and blood pharmacokinetics of iodine I 131 monoclonal antibody 3F8 and serum human antimouse antibodies. Samples are also analyzed in tumor genetic studies.

After completion of study treatment, patients are followed periodically for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of a malignancy known to expressGD2. Such tumors include medulloblastoma/primitive neuroectodermal tumor of the CNS, high grade astrocytomas, malignant glioma, neuroblastoma, retinoblastoma, ependymoma, rhabdoid tumors, sarcomas, melanoma or small cell lung carcinoma. For patients with other tumor types, GD2 expression must be confirmed by immunohistochemical staining and assessed by the Department of Pathology using prior frozen tissue, bone marrow or CSF cytology (send to Research Lab).
* Patients must have CNS/ leptomeningeal disease including high risk medulloblastoma, or a CNS/leptomeningeal malignancy which is refractory to conventional therapies, or for which no conventional therapy exists, OR a recurrent brain tumors with a predilection for leptomeningeal dissemination (medulloblastoma, PNET, rhabdoid tumor).
* Patients must have an absolute neutrophil count (ANC) > 1000/ul and a platelet count > 50,000/ul.
* Patients may have active malignancy outside the central nervous system.
* Patients who have a programmable shunt will not be excluded.
* Both pediatric and adult patients of any age are eligible.
* Patients or a legal guardian will sign an informed consent form approved by the IRB and obtained by the Principal or a Co- Investigator before patient entry. Minors will provide assent.

Exclusion Criteria:

* Patients with obstructive or symptomatic communicating hydrocephalus.
* Patients with an uncontrolled life-threatening infection.
* Patients who are pregnant: Pregnant women are excluded for fear of danger to the fetus. Therefore negative pregnancy test is required for all women of child-bearing age, and appropriate contraception is required during the study period.
* Patients who have received cranial or spinal irradiation less than 3 weeks prior to the start of this protocol.
* Patients who have received systemic chemotherapy (corticosteroids not included) less than 3 weeks prior to the start of this protocol.
* Severe major organ toxicity. Specifically, renal, cardiac, hepatic, pulmonary, and gastrointestinal system toxicity should all be less than or equal to grade 2. Patients with stable neurological deficits (because of their brain tumor) are not excluded. Patients with <= 3 hearing loss are not excluded.
* Patients must have no rapidly progressing or deteriorating neurologic examination.
* Patients who have already received >45 Gy to the craniospinal radiation or >72 Gy focal brain radiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Kramer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 131I-3F8: This is a phase II single-arm open-label study that will define responses to therapy with weekly intrathecal 131I-3F8 in patients with central nervous system/leptomeningeal GD2-expressing disease.
  DNA analysis
  immunologic technique
  pharmacological study
  iodine I 131 monoclonal antibody 3F8
  131I-3F8: Patients will receive 10mCi intrathecal 131I-3F8 per week. Patients will be pre-medicated with dexamethasone to prevent possible meningeal inflammatory reaction, Liothyronine and SSKI to prevent thyroid accumulation, and acetaminophen and diphenhydramine in anticipation of possible allergic reaction and fever.
Period: Overall Study
Arm/Group | 131I-3F8
Started | 78
Completed | 45
Not Completed | 33
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Enrolled but not treated | 1
Not completed — Removed due to progressive disease | 29

BASELINE CHARACTERISTICS:
Arm/Group | 131I-3F8
Number analyzed (Participants) | 78
Age, Continuous [Mean (Full Range); unit: years] | 10 [1 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 63
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Six-month Overall Survival
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 131I-3F8
Number analyzed (Participants) | 78
Participants
  Participants still alive at the 6-month mark | 67
  Participants not alive at the 6-month mark | 11

2. Primary Outcome: Number of Participants With Response at 6 Months
Description: Complete Response (CR): Cytologic and radiographic CR will be evaluated separately, since patients with cytologic clearing and clinical response may continue to have residual abnormalities on MRI scans. Patients with a CR must also have stable or improved neurologic exam.
  Stable Disease (SD): Exists when a patient fails to fulfill the criteria for either complete or partial response or progressive disease.
  Progressive Disease (PD): An increase of at least 50% in the absolute number of malignant cells in the CSF OR, in -solid tumor patients, an increase of greater than 25% in the size of measurable lesions on MR scan OR the recurrence of malignant cells in the CSF or new lesions on MR after a patient has attained a complete remission OR evidence of clinical neurologic progression. New sites of or increasing evidence of leptomeningeal enhancement that is not "measurable" will also be considered evidence of disease progression.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 131I-3F8
Number analyzed (Participants) | 78
Participants
  Complete Response | 31
  Stable Disease | 8
  Progression of Disease | 21
  Not Evaluable | 18

3. Secondary Outcome: Number of Participants Evaluable for Toxicities
Description: Toxicities will be assessed via the NCI toxicity criteria (CTC 3.0).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 131I-3F8
Number analyzed (Participants) | 78
Participants
  Evaluable for toxicities | 77
  Not evaluable for toxicities, participant was not treated | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 131I-3F8
All-Cause Mortality (participants affected / at risk) | 54/78
Serious Adverse Events (participants affected / at risk) | 39/78
Other Adverse Events (participants affected / at risk) | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 131I-3F8 (N=78)
ALT, SGPT (Investigations) | 1
Bilirubin (Investigations) | 1
Confusion (Psychiatric disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 6
Gastrointestinal, other (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 2
Inf norm ANC/gr1/2 neut- (Infections and infestations) | 2
Infection, other (Infections and infestations) | 3
Injection site reaction/extravasation (Injury, poisoning and procedural complications) | 1
Lipase (Investigations) | 1
Lymphopenia (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Nerology - Other (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Pain - bone (Musculoskeletal and connective tissue disorders) | 1
Pain - Head/headache (Nervous system disorders) | 5
Pain - other (General disorders) | 2
Platelets (Investigations) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Psychosis (Psychiatric disorders) | 1
Seizure (Nervous system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Somnolence (Nervous system disorders) | 2
Vision-blurred vision (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 131I-3F8 (N=78)
Hypoalbuminemia (Metabolism and nutrition disorders) | 26
Alkaline phosphatase (Investigations) | 8
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
ALT, SGPT (Investigations) | 63
Amylase (Investigations) | 3
AST, SGOT (Investigations) | 55
Bicarbonate, serum-low (Investigations) | 1
Hyperbilirubinemia (Investigations) | 10
Hypercalcemia (Metabolism and nutrition disorders) | 4
Cholesterol high (Investigations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 77
Hypoglycemia (Metabolism and nutrition disorders) | 15
Hemoglobin (Blood and lymphatic system disorders) | 77
Hypertension (Vascular disorders) | 3
INR (Investigations) | 11
Leukocytes (Investigations) | 77
Lymphopenia (Investigations) | 77
Hypomagnesemia (Metabolism and nutrition disorders) | 13
Muscle weakness - Extremity - lower (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Neutrophils/granulocytes (Investigations) | 77
Pain - head/headache (Nervous system disorders) | 3
Platelets (Investigations) | 77
Hyperkalemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 42
PTT (Investigations) | 15
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 21
Tremor (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Somnolence (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 13
Pain (General disorders) | 1
Lipase (Investigations) | 2
Hypotension (Vascular disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Gastrointestinal, other (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT00445965/Prot_SAP_000.pdf